CLINICAL TRIAL: NCT04675333
Title: A Phase 2 Study of ALX148 in Combination With Pembrolizumab and Chemotherapy in Patients With Advanced Head and Neck Squamous Cell Carcinoma (ASPEN-04)
Brief Title: Evorpacept (ALX148) in Combination With Pembrolizumab and Chemotherapy in Patients With Advanced Head and Neck Squamous Cell Carcinoma (ASPEN-04)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ALX Oncology Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT148004; KEYNOTE-B88 (Other: Merck Sharp & Dohme LLC); MK-3475-B88 (Other: Merck Sharp & Dohme LLC); 2020-004662-19 (EudraCT Number); 2023-508342-17-00 (EU CTIS Number)
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: ALX148; CD47; SIRPα; HNSCC; pembrolizumab; evorpacept
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — ALX148; pembrolizumab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- evorpacept (ALX148) + pembrolizumab + Chemotherapy (Experimental): evorpacept (ALX148) 45 mg/kg IV, pembrolizumab 200 mg IV, and chemotherapy given every 3 weeks.
  Interventions: Drug: evorpacept; Drug: pembrolizumab; Drug: Cisplatin/Carboplatin; 5FU
- pembrolizumab + Chemotherapy (Active Comparator): pembrolizumab 200 mg IV and chemotherapy given every 3 weeks.
  Interventions: Drug: pembrolizumab; Drug: Cisplatin/Carboplatin; 5FU

INTERVENTIONS:
Drug: evorpacept — IV Q3W
  Other Names: ALX148
  Arms: evorpacept (ALX148) + pembrolizumab + Chemotherapy
Drug: pembrolizumab — IV Q3W
  Other Names: KEYTRUDA®
Drug: Cisplatin/Carboplatin; 5FU — IV Q3W
  Other Names: Platinol/Paraplatin; Adrucil

SUMMARY:
A Phase 2 Study of evorpacept (ALX148) in Combination With pembrolizumab and Chemotherapy in Patients With Advanced Head and Neck Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
This is a open-label, randomized phase 2 multi-center study of the anti-tumor efficacy of evorpacept (ALX148) + pembrolizumab + 5FU + platinum and of pembrolizumab + 5FU + platinum in patients with metastatic or unresectable, recurrent HNSCC who have not yet been treated for their advanced disease. The study comprises of an initial safety lead-in followed by a randomized portion.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated metastatic or unresectable, recurrent head and neck squamous cell carcinoma.
* Adequate bone marrow function.
* Adequate renal and liver function.
* Adequate ECOG performance status.

Exclusion Criteria:

* Patients with known symptomatic CNS metastases or leptomeningeal disease requiring steroids.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Prior treatment with any anti-CD47 or anti-SIRPα agent.
* Prior treatment with anti-PD-1 or PD-L1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate per RECIST 1.1 | Last randomized patient reaching at least 24 weeks of follow-up

SECONDARY OUTCOMES:
Duration of response | Up to 36 months
Progression-free survival | Up to 36 months
Overall survival | Up to 36 months
Adverse events | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (44):
- United States (13):
  - Hoag Hospital, Irvine, California
  - University of California San Diego, La Jolla, California
  - Cedar Sinai Medical Center, Los Angeles, California
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical System, Baltimore, Maryland
  - Memorial Sloan Kettering, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University/ Knight Cancer Institute, Portland, Oregon
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist Cancer Center, Houston, Texas
- Australia (4):
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Ashford Cancer Centre, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Groeninge, Kortrijk
- Netherlands (2):
  - Amsterdam UMC, Locatie VUMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- Singapore (2):
  - National University Cancer Institute, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju-si
  - Yeungnam University Medical Center, Daegu
  - Gachon University (GCU) - Gil Medical Center (Gil Hospital), Incheon
  - Seoul National University, Bundang Hospital, Seongnam
  - CHA University - Bundang CHA General Hospital (CHA Bundang Medical Center), Seongnam-si
  - The Catholic University of Korea - Eunpyeong St. Mary's Hospital, Seoul
  - Seoul National University Hospital (SNUH) - SMG-SNU Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Universitari Dexeus, Barcelona, Barcelona
  - Institut Catala d Oncologia (ICO), Badalona
  - Institut Catala dOncologia, L'Hospitalet de Llobregat
  - Hospital Universitario Severo Ochoa, Leganés
  - Grupo Hospital de Madrid (HM) - Hospital Universitario Madrid Sanchinarro - Cent, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario de Navarra, Pamplona
- United Kingdom (3):
  - The Royal Marsden Hospital - Surrey, London
  - University College London Hospital, London
  - The Royal Marsden Hospital- London, London

IPD SHARING:
Plan to Share IPD: No